CLINICAL TRIAL: NCT03565666
Title: The Insulin-Only Bionic Pancreas Bridging Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Clinical Study Director, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000853
Record Dates: First submitted 2018-05-29; First posted 2018-06-21 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Type1 Diabetes Mellitus
Keywords: bionic pancreas; closed loop; insulin; continuous glucose monitor
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Adult RCT: Usual care (Active Comparator): Participants randomized to usual care first started the usual care arm (UC) managing their diabetes with either multiple daily injections or continuous subcutaneous insulin infusion (pump therapy) for 7 days. All subjects wore a Dexcom G5 continuous glucose monitor (CGM) and half of all subjects also were a senseonics CGM. The usual care period was followed by the other 2 arms according to each subject's randomization schedule
  Interventions: Other: Usual care
- Adult RCT: closed-loop control with iLet Humalog or Novolog (Experimental): Participants randomized to the iLet with humalog/novolog first started the insulin-only iLet arm using the insulin analog that they use for their usual care (either Humalog or Novolog). All subjects wore a Dexcom G5 CGM and half of all subjects also wore a Senseonics Eversense CGM. The iLet period was followed by the other 2 arms according to each subject's randomization schedule
  Interventions: Device: iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog
- Adult RCT: closed-loop control with iLet using Fiasp (Experimental): Participants randomized to the iLet with Fiasp first started the insulin-only iLet arm using faster insulin aspart (Fiasp) in PumpCart, where the pharmacokinetic (PK) parameter for tmax used by the insulin-dosing algorithm was set to the same value as is used for Humalog and Novolog (65 minutes). All subjects wore a Dexcom G5 CGM and half of all subjects also wore a Senseonics Eversense CGM. The iLet period was followed by the other 2 arms according to each subject's randomization schedule
  Interventions: Drug: iLet Bionic Pancreas insulin-only configuration with Fiasp

INTERVENTIONS:
Device: iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog — iLet Bionic Pancreas insulin-only configuration with Humalog or Novolog
  Arms: Adult RCT: closed-loop control with iLet Humalog or Novolog
Drug: iLet Bionic Pancreas insulin-only configuration with Fiasp — iLet Bionic Pancreas insulin-only configuration with Fiasp (faster insulin aspart)
  Arms: Adult RCT: closed-loop control with iLet using Fiasp
Other: Usual care — Usual care
  Arms: Adult RCT: Usual care

SUMMARY:
The iLet is a closed-loop delivery system that can be used in insulin-only, bihormonal, or glucagon-only configurations. Previous studies have utilized a phone-based bionic pancreas. The iLet consists of a touchscreen-enabled, menu-driven user interface and an onboard microprocessor that provides a comprehensive and standalone platform, which allows the iLet to operate independently of smartphones or other devices and without the need for internet support during routine operation.

This is a multicenter study of adult participants with type 1 diabetes, who will manage their diabetes with the iLet bionic pancreas compared to usual care.

DETAILED DESCRIPTION:
This study will serve as a transitional study, bridging to larger and longer outpatient pivotal studies using the insulin-only configuration of the bionic pancreas.

The Adult RCT Period will consist of a multi-center, three-period, random-order, cross-over, feasibility study in 36 adult participants ≥ 18 years old with T1D. Insulin therapy for each participant will be administered (i) using the iLet in the insulin-only configuration and the insulin analog that they use for their usual care (either Humalog or Novolog) for 7 days, (ii) in another period using the iLet in the insulin-only configuration with faster insulin aspart (Fiasp) for 7 days (iii) in a third period using the participant's own usual care (UC) for 7 days. All three experimental periods will be followed by round-the-clock, remote, telemetric monitoring for hyperglycemia (> 300 mg/dl for ≥ 90 minutes) and hypoglycemia (< 50 mg/dl for ≥ 15 minutes). Half the subjects enrolled were expected to manage their diabetes with MDI and the other half with insulin pumps in their UC. An implantable Eversense CGM will also be placed in half the study participants for a CGM comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Diabetes managed using an insulin pump for ≥ 3 months or with multiple daily injections (approximately 1/2 of participants should use a pump and approximately 1/2 should use MDI)
3. Age ≥18 years;

   • There is no upper age limit in the Adult RCT Period (instead the exclusion criteria are used to restrict the participants to those healthy enough to participate in the trial)
4. HbA1c level <11.0%

   • A point of care or local lab measurement is used to assess eligibility for screening.
5. At least 3 SMBG meter tests daily on average or use of a CGM and 2 or more SMBG meter tests daily on average by history
6. For females, not currently known to be pregnant

   • If female, sexually active, and at risk for pregnancy, must agree to use a highly effective form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all women who are post-menarche and pre-menopause who are not surgically sterile. Participants who become pregnant will be discontinued from the study.
7. An understanding of and willingness to follow the protocol and sign the informed consent and assent where applicable

Exclusion Criteria:

-The presence of any of the following is an exclusion for the study:

1. Unable to provide informed consent (e.g. impaired cognition or judgment)
2. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the BP, impaired memory)
3. Unable to speak and read English
4. Currently using for the first time a real-time CGM for < 1 month (Individuals who have been using CGM for 1 or more months are eligible)
5. Current use of non-FDA approved closed-loop or hybrid closed-loop insulin delivery system
6. Current use of insulin glulisine (Apidra) as part of usual diabetes home regimen
7. Current off-label use of faster-acting insulin aspart (Fiasp) in CSII therapy as part of usual diabetes home regimen
8. Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the participant
9. Pregnant (positive urine HCG), breast feeding, plan to become pregnant in the next 12 months, or sexually active and at risk for pregnancy without use of contraception
10. Current alcohol abuse (intake averaging >4 drinks daily in last 30 days) or other substance abuse (use within the last 3 months of controlled substances other than marijuana without a prescription)
11. Unwilling or unable or to avoid use of drugs that may dull the sensorium, reduce sensitivity to symptoms of hypoglycemia, or hinder decision making during the period of participation in the study (use of benzodiazepines or narcotics, even if by prescription, may be excluded according to the judgment of the principal investigator)
12. Stage 4 renal failure (eGFR <30) or Stage 5 renal failure on dialysis (hemodialysis or peritoneal dialysis)
13. History of cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
14. Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. exercise of intensity up to 6 METS) despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
15. Abnormal EKG consistent with increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, proximal LAD critical stenosis (Wellen's sign), or prolonged QT interval (> 440 ms). Other EKG findings, including stable Q waves, are not grounds for exclusion as long as the participant is not excluded according to other criteria. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.

    • EKG is only required for participants ≥50 years old or with diabetes duration ≥20 years
16. For participants < 50 years of age and < 20 years since diagnosis: History of prolonged QT interval, malignant arrhythmia, or congenital heart disease
17. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV
18. History of TIA or stroke in the last 12 months
19. Recent history of diabetic ketoacidosis (DKA) or severe hypoglycemia in the last 6 months. Severe hypoglycemia is defined as an event that required assistance of another person due to altered consciousness, and required another person to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or coma.
20. History of more than 1 episode of DKA requiring hospitalization in the last 2 years
21. History of more than 1 episode of severe hypoglycemia in the last year.
22. Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with anti-psychotic medications that are known to affect glucose regulation.
23. Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference
24. Unable or unwilling to completely avoid acetaminophen for duration of study
25. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
26. History of eating disorder within the last 2 years, such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
27. Current or planned use of SGLT2 inhibitors (prior use more than 3 months prior to enrollment is acceptable; SGLT2 inhibitors should not be initiated during the trial)
28. If using GLP1, pramlintide, or metformin must be on a stable dose for 3 months prior to enrollment (these agents should not be initiated during the trial)
29. Required use of 2 or more steroid bursts in the 6 months prior to the trial
30. History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
31. Any factors that, in the opinion of the site principal investigator or clinical protocol chair, would interfere with the safe completion of the study, including medical conditions that may require hospitalization during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Nemours Children's Specialty Care, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be published as online supplemental material to the main paper describing the results, as we have done for all of our previous bionic pancreas studies.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 participants were recruited at MGH and 18 participants at Stanford
Pre-assignment Details: This study consisted of a test-run period followed by an RCT
Groups:
- Usual Care Then Either iLet/Novolog/Humalog or iLet/Fiasp: Participants first started the usual care arm (managing their diabetes with either multiple daily injections or insulin pump) for 7 days, then switched to either the insulin-only iLet using Novolog or Humalog for 7 days, or the insulin-only iLet using Fiasp for 7 days. No washout period was required between arms
- iLet/Novolog/Humalog Then Either iLet/Fiasp or Usual Care: Participants first started using the insulin-only iLet with either Novolog or Humalog for 7 days then switched to either the usual care arm (managing their diabetes with multiple daily injections or insulin pump) for 7 days, or the insulin-only iLet arm using Fiasp for 7 days. No washout period was required between arms.
- iLet/Fiasp Then Either iLet With Novolog/Humalog or Usual Care: Participants first started the insulin-only iLet using Fiasp for 7 days, then switched to either the insulin-only iLet arm using Novolog or Humalog for 7 days or the usual care arm, (managing their diabetes with either multiple daily injections or insulin pump) for 7 days. No washout period was required between arms
Period: Overall Study
Arm/Group | Usual Care Then Either iLet/Novolog/Humalog or iLet/Fiasp | iLet/Novolog/Humalog Then Either iLet/Fiasp or Usual Care | iLet/Fiasp Then Either iLet With Novolog/Humalog or Usual Care
Started | 12 | 12 | 12
Completed | 12 | 12 | 11
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 36 adult patients with type 1 diabetes will complete 3 arms in a random-order crossover fashion. Participants in the usual care arm (UC) will manage their diabetes with either multiple daily injections or continuous subcutaneous insulin infusion (pump therapy). All subjects will wear Dexcom G5 continuous glucose monitor (CGM) and half of all subjects will also wear a senseonics CGM.
  Each arm is 7 days, no washout between arms
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant was not analysed as they discontinued the study after 1 day and did not meet the criteria for their results to be included in the analyses (according to the protocol)
  Participants
    number analyzed (Participants) | 35
    <=18 years | 0
    Between 18 and 65 years | 32
    >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-hispanic | 28
  Bklack/African-American | 1
  Asian | 5
  American Indian/Alaskan Native | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: 1 participant was not analysed as they discontinued the study after 1 day and did not meet the criteria for their results to be included in the analyses (according to the protocol)
  Participants
    United States: number analyzed (Participants) | 35
    United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean CGM Glucose
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Usual Care Arm: Participants who completed 7 days of managing their diabetes with their usual care (either MDI or insulin pump) during the 3 weeks of the study period 35 participants completed this arm
- iLet With Insulin Analogue (Novolog/Humalog) Arm: Participants who completed 7 days of using the iLet with either Novolog or Humalog to manage their diabetes during the 3 weeks of the study period 34 participants completed this arm
- iLet Using Fiasp Arm: Participants who completed 7 days of using the iLet with faster acting aspart (Fiasp) to manage their diabetes during the 3 weeks of the study period 35 participants completed this arm
Arm/Group | Usual Care Arm | iLet With Insulin Analogue (Novolog/Humalog) Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
mg/dl | 144.3 (9.5) | 162 (26) | 155 (12)

2. Primary Outcome: Percentage of Time Where Glucose is Less Than 54 mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Usual Care Arm | iLet With Insulin Analogue (Novolog/Humalog) Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 0.58 [0.39 to 0.93] | 0.53 [0.18 to 0.98] | 0.56 [0.17 to 1.12]

3. Other Pre Specified Outcome: Episodes of Severe Hypoglycemia
Description: Pre-specified to report the total number of episodes summed across all participants
Time Frame: Days 3-7 for the RCT Period
Measure: Number; unit: number of episodes
Arm/Group | Usual Care Arm | iLet With Insulin Analogue (Novolog/Humalog) Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 36
number of episodes | 0 | 0 | 1

4. Other Pre Specified Outcome: Episodes of Diabetic Ketoacidosis (DKA)
Description: pre-specified to report the total number of episodes summed across all participants
Time Frame: Days 3-7 for the RCT Period
Measure: Number; unit: number of episodes
Arm/Group | Usual Care Arm | iLet With Insulin Analogue (Novolog/Humalog) Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
number of episodes | 0 | 0 | 0

5. Other Pre Specified Outcome: Percentage of Time Where Glucose is Less Than 70 mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- iLet Using Humalog/Novolog Arm: Participants who completed 7 days of using the iLet with either Novolog or Humalog to manage their diabetes during the 3 weeks of the study period 34 participants completed this arm
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 5.09 [3.73 to 5.5] | 3.2 [1.3 to 5.2] | 2.7 [1.5 to 3.9]

6. Other Pre Specified Outcome: Percentage of Time in the Glucose Target Range of 70-180 mg/dl
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 73.3 (7.35) | 62.2 (16.2) | 69.2 (9.2)

7. Other Pre Specified Outcome: Percentage of Time Where Glucose is Greater Than 180 mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 21.8 (7.6) | 34.4 (16.9) | 27.96 (8.9)

8. Other Pre Specified Outcome: Percentage of Time Where Glucose is Less Than 60 mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 1.67 (0.73) | 1.3 (1.23) | 1.19 (0.93)

9. Other Pre Specified Outcome: Percentage of Time Where Glucose is Greater Than 250 mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 3.64 (3.03) | 10.42 (10.43) | 7.73 (4.99)

10. Other Pre Specified Outcome: Percentage Time in the Glucose Target Range of 70-120mg/dL
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Usual Care Arm | iLet Using Humalog/Novolog Arm | iLet Using Fiasp Arm
Number analyzed (Participants) | 35 | 34 | 35
percentage of time | 30.65 (4.17) | 25.65 (12.36) | 28.24 (7.98)

11. Other Pre Specified Outcome: Mean Absolute Relative Difference Between Dexcom G5 CGM and Contour Next One Glucose Meter
Description: The MARD is calculated as the mean value of individual absolute relative differences (ARD). The ARD is calculated as follows: 100*(CGM-reference glucose)/reference glucose
Time Frame: Days 3-7 for the RCT Period
Measure: Mean (Standard Deviation); unit: MARD (CGMG-meter glucose)/meter glucose)
Groups:
- RCT Period Days 1-7: 36 adult patients with type 1 diabetes will complete 3 arms in a random-order crossover fashion. Half of the subjects (n=18) will wear the Dexcom G5 continuous glucose monitor (CGM) and the other half will wear a Senseonics Eversense CGM.
Arm/Group | RCT Period Days 1-7
Number analyzed (Participants) | 18
MARD (CGMG-meter glucose)/meter glucose) | 18.8 (8.2)

12. Other Pre Specified Outcome: Mean Absolute Relative Difference Between Senseonics Eversense CGM and Contour Next One Glucose Meter
Description: as for outcome 11
Time Frame: Days 1-7 of the Adult RCT period
Measure: Mean (Standard Deviation); unit: MARD: Mean of all [(CGMG - PG)/PG]
Groups:
- Days 1-7 of RCT: 36 adult patients with type 1 diabetes will complete 3 arms in a random-order crossover fashion. Half of the subjects (n=18) will wear the Dexcom G5 continuous glucose monitor (CGM) and the other half will wear a Senseonics Eversense CGM.
Arm/Group | Days 1-7 of RCT
Number analyzed (Participants) | 18
MARD: Mean of all [(CGMG - PG)/PG] | 13.3 (5)

ADVERSE EVENTS:
Time Frame: Up to 2 months for the RCT
Groups:
- Usual Care Arm: Participants who completed 7 days of managing their diabetes with their usual care (either MDI or insulin pump) during the 3 weeks of the study period 35 participants completed this arm
  Usual care: Usual care
- iLet With Humalog/Novolog Arm: Participants who completed 7 days of using the iLet with either Novolog or Humalog to manage their diabetes during the 3 weeks of the study period 34 participants completed this arm
Arm/Group | Usual Care Arm | iLet With Humalog/Novolog Arm | iLet Using Fiasp Arm
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 1/36
Other Adverse Events (participants affected / at risk) | 4/36 | 15/36 | 16/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Arm (N=36) | iLet With Humalog/Novolog Arm (N=36) | iLet Using Fiasp Arm (N=36)
Serious adverse event (Endocrine disorders) | 0 | 0 | 1 (1) — Severe hypoglycemia defined as hypoglycemia necessitating the aid of a third party for recovery
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Arm (N=36) | iLet With Humalog/Novolog Arm (N=36) | iLet Using Fiasp Arm (N=36)
Non-serious adverse event (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) — Elevated ketones >1.0 mmol/L (no DKA)
Non serious adverse event (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — Nausea without vomiting
Non-serious adverse event (Endocrine disorders) | 4 (10) | 14 (19) | 15 (27) — Hypoglycemia For the test run, data for hypos is collected from RedCap surveys and for RCT data is collected from CGM downloads

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT03565666/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03565666/SAP_001.pdf